CLINICAL TRIAL: NCT04924569
Title: Continence Care Registry (ConCaRe™)
Brief Title: Continence Care Registry
Acronym: ConCaRe™
Status: Active, not recruiting | Type: Observational
Sponsor: Hollister Incorporated (Industry)
Collaborators: Parexel (Industry); Technomics Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 6016-CONT
Record Dates: First submitted 2021-05-31; First posted 2021-06-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Neurogenic Bladder; Non-Neurogenic Bladder
Keywords: Intermittent Self Catheterization; Intermittent catheter; Urinary retention; Urinary incontinence; Urinary symptoms; Urinary tract infection (UTI)
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention; Urinary Incontinence; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care: Individuals using an intermittent catheter to void urine through the urethra. Participants use their currently prescribed intermittent catheter per their clinician's standard of care.

SUMMARY:
This observational research study aims to build a multinational electronic patient-reported outcomes (ePRO) registry of adult end users in outpatient and community settings using intermittent catheter(s) to void via the urethra to manage urinary retention and incomplete bladder emptying. Research participants will be asked to self-report on various attributes of their currently prescribed intermittent catheters and other various aspects of using an intermittent catheter.

DETAILED DESCRIPTION:
This observational research study aims to build a multinational ePRO registry of adult end users in outpatient and community settings using intermittent catheter(s) to void via the urethra to manage urinary retention and incomplete bladder emptying. Research resulting from data generated from an ePRO registry will factor in end user perspectives on intermittent catheterization habits and behaviors and intermittent catheter performance to inform and guide healthcare providers, end users, and caregivers in making the most informed healthcare decisions regarding intermittent catheterization. Research participants will be asked to self-report on various attributes of their currently prescribed intermittent catheters and various aspects of habits and behaviors, including health-related quality of life, of using an intermittent catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age; male or female.
2. Is performing transurethral intermittent catheterization.
3. Uses intermittent catheter(s) from any manufacturer as a form of management for urinary retention or incomplete bladder emptying.
4. Must be able to provide informed consent and have no cognitive impairment that would hinder the ability to provide informed consent or self-reported data.
5. Lives and has permanent residence in one of the countries that the study is being conducted at time of enrollment (USA, Canada, UK, Germany, France, The Netherlands, or Italy)
6. Is willing and able to complete electronic questionnaires monthly for the first year of data collection and quarterly thereafter or appoint a caregiver proxy.
7. Is able to read and respond to the questionnaires in the language options provided for a given country (e.g. French Canadian or English for Canada)

Exclusion Criteria:

1. Performs non transurethral catheterization, e.g., stoma.
2. Participating in a clinical study involving transurethral intermittent self-catheterization at the time of enrollment.
3. Employee of Sponsor at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sponsor-curated customer databases and printed EC/IRB approved advertisements targeted to intermittent catheter consumers from the USA, Canada, UK, Italy, France, Germany, and The Netherlands that may be distributed by clinicians, mail, website, conferences and other consumer contacts.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Creation of longitudinal continence care ePRO-based, direct-to-consumer registry | 5 years
  To build a longitudinal continence care ePRO-based, direct-to-consumer registry addressing overall intermittent self-catheterization product satisfaction, QoL, healthcare resource utilization associated with urinary symptoms, urinary tract infections and other complications including burden of ISC over time, and end-user product preference factors.

SECONDARY OUTCOMES:
Identification of intermittent self-catheterization habits and behaviors | 5 years
  To identify intermittent self-catheterization habits and behaviors, and enable meaningful intermittent catheter comparisons, including but not limited to product-specific outcomes related to urinary symptoms associated with ISC, frequency of UTI and other complications over time, and product satisfaction over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Simmons, DNP, APRN, FNP-C, CWON, DNC, Principal Investigator — Hollister Incorporated; Diane Newman, D.N.P. F.A.A.N. B.C.B.-P.M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hollister Incorporated, Libertyville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] New PW. The evidence supporting single-use intermittent catheters in people with spinal cord injury. Spinal Cord Ser Cases. 2020 Sep 30;6(1):89. doi: 10.1038/s41394-020-00339-5. PMID 32999268
- [Background] Romo PGB, Smith CP, Cox A, Averbeck MA, Dowling C, Beckford C, Manohar P, Duran S, Cameron AP. Non-surgical urologic management of neurogenic bladder after spinal cord injury. World J Urol. 2018 Oct;36(10):1555-1568. doi: 10.1007/s00345-018-2419-z. Epub 2018 Jul 26. PMID 30051263
- [Background] Letica-Kriegel AS, Salmasian H, Vawdrey DK, Youngerman BE, Green RA, Furuya EY, Calfee DP, Perotte R. Identifying the risk factors for catheter-associated urinary tract infections: a large cross-sectional study of six hospitals. BMJ Open. 2019 Feb 21;9(2):e022137. doi: 10.1136/bmjopen-2018-022137. PMID 30796114
- [Background] Kinnear N, Barnett D, O'Callaghan M, Horsell K, Gani J, Hennessey D. The impact of catheter-based bladder drainage method on urinary tract infection risk in spinal cord injury and neurogenic bladder: A systematic review. Neurourol Urodyn. 2020 Feb;39(2):854-862. doi: 10.1002/nau.24253. Epub 2019 Dec 17. PMID 31845396
- [Background] Newman DK, New PW, Heriseanu R, Petronis S, Hakansson J, Hakansson MA, Lee BB. Intermittent catheterization with single- or multiple-reuse catheters: clinical study on safety and impact on quality of life. Int Urol Nephrol. 2020 Aug;52(8):1443-1451. doi: 10.1007/s11255-020-02435-9. Epub 2020 Mar 14. PMID 32172456
- [Background] Rognoni C, Tarricone R. Intermittent catheterisation with hydrophilic and non-hydrophilic urinary catheters: systematic literature review and meta-analyses. BMC Urol. 2017 Jan 10;17(1):4. doi: 10.1186/s12894-016-0191-1. PMID 28073354
- [Background] Logan, K. Intermittent self-catheterisation in men. Trends Urology & Men Health, 2018;9: 11-14.
- [Background] International Organization for Standardization. Clinical investigation of medical devices for human subjects-Good clinical practice 2011;ISO 14155.
- [Background] ISPE. Guidelines for good pharmacoepidemiology practices (GPP). Pharmacoepidemiol Drug Saf. 2008 Feb;17(2):200-8. doi: 10.1002/pds.1471. No abstract available. PMID 17868186